CLINICAL TRIAL: NCT02264249
Title: Residual Gastric Volume in Same Day Versus Split Dose and Evening Before Bowel Preparation: A Prospective Observational Study
Brief Title: Residual Gastric Volume in Same Day Versus Split Dose and Evening Before Bowel Preparation
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Alison Schneider, Staff Physician, The Cleveland Clinic
Other Study IDs: FLA 14-086
Record Dates: First submitted 2014-10-06; First posted 2014-10-15 (Estimated); Results first posted 2016-09-09 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Esophagogastroduodenoscopy; Colonoscopy
MeSH Terms: interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Split dose colonoscopy preparation: Esophagogastroduodenoscopy and colonoscopy - split dose - ½ evening before and ½ early AM (4L volume or 2L volume bowel preparation)
  Interventions: Other: Esophagogastroduodenoscopy and colonoscopy split dose prep
- Evening before colonoscopy preparation: Esophagogastroduodenoscopy and colonoscopy - Evening before (4L, 2L or miralax bowel preparation)
  Interventions: Other: Esophagogastroduodenoscopy and colonoscopy Evening before colonoscopy prep
- Same day prep colonoscopy preparation: Esophagogastroduodenoscopy and colonoscopy - Same day prep (4L volume or 2L volume or Miralax bowel preparation)
  Interventions: Other: Esophagogastroduodenoscopy and colonoscopy Same day prep colonoscopy preparation

INTERVENTIONS:
Other: Esophagogastroduodenoscopy and colonoscopy split dose prep — Patients undergoing a combined EGD (esophagogastroduodenoscopy) and a colonoscopy receive the Split dose colonoscopy prep
  split dose colonoscopy preparation- ½ evening before and ½ early AM (4L volume or 2L volume bowel preparation)
  Groups: Split dose colonoscopy preparation
Other: Esophagogastroduodenoscopy and colonoscopy Evening before colonoscopy prep — Patients undergoing a combined EGD (esophagogastroduodenoscopy) and a colonoscopy receive Evening before (4L, 2L or miralax bowel preparation)
  Groups: Evening before colonoscopy preparation
Other: Esophagogastroduodenoscopy and colonoscopy Same day prep colonoscopy preparation — Patients undergoing a combined EGD (esophagogastroduodenoscopy) and a colonoscopy receive Same day prep (4L volume or 2L volume or Miralax bowel preparation)
  Groups: Same day prep colonoscopy preparation

SUMMARY:
The purpose of this study is to determine residual gastric volume and residual gastric pH in patients undergoing combined EGD and colonoscopy comparing the standard single dose prep with the split dose bowel preparation and same day bowel preparations.

DETAILED DESCRIPTION:
The ASGE and ACG have developed standards for high-quality colonoscopy and ADR. Bowel cleansing must be optimal to enhance polyp detection and several studies have demonstrated the advantage of split dose or same day preparation as opposed to ingesting the preparation the day before. It is recommended that patients undergo split dosing of the bowel preparation or even same day bowel preparation for optimal cleansing. This is critical for high quality colonoscopy.

One of the risks associated with colonoscopy is pulmonary aspiration. Part of this risk may be related to retained gastric volume and gastric pH at the time of the endoscopic procedures. Aspiration pneumonia may be related to the acidity where more acidic aspirate may cause more severe respiratory compromise. In a recent article, Huffman supported the safety of split dose bowel preparation (4L bowel preparation) for outpatients undergoing colonoscopy. In this study it was/found that residual gastric volume in split dose preparations was higher than patients undergoing EGD alone but was not different from than in patients receiving bowel preparation the evening before. Early morning bowel preps for patients undergoing upper and lower endoscopies was not evaluated in this study. To our knowledge, the relationship of residual gastric volume in same day bowel preps has not been evaluated and has not been compared with the split dose bowel preps. A formal evaluation of difference in gastric acidity has not been evaluated in patients undergoing bowel prep for colonoscopy.

The study has a prospective observational design. The patients who have been already scheduled for a combined esophagogastroduodenoscopy and colonoscopy for their specific indications will be asked to be a part of this study. No additional intervention will be done other than the procedure they were already scheduled for. No specific interventions will be assigned to the subjects of the study. Outcomes will be assessed in pre-defined groups based on the bowel preparation taken by the patient.

The fluid is going to be collected in a suction container without solidifier material. Once the endoscopist enters the stomach all fluid will be suctioned which is part of the customary process of endoscopy. Once all fluid is aspirated, the container will be removed to empty the fluid into a measuring canister while the endoscopic procedure is continued and a container with solidifier material is instead connected to suction. The pH will be measured on the gastric fluid that was aspirated using a calibrated catheter pH device.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (ages 18 and over) scheduled for elective non-emergency outpatient combined Esophagogastroduodenoscopy and colonoscopy procedures at CCF. No additional intervention will be done other than the procedure they were scheduled for.

Exclusion Criteria:

1. Upper GI or lower GI bleeding at the time of procedure
2. Large amounts of vomiting reported before the procedure (with bowel preparation)
3. Hospital inpatients
4. History of abdominal surgery
5. History of gastroparesis or other documented GI transit disorder (ex. Colonic inertia)
6. Pregnancy Patients with diabetes mellitus taking Metoclopramide without proven gastroparesis by formal testing will not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (ages 18 and over) scheduled for elective non-emergency outpatient combined Esophagogastroduodenoscopy and colonoscopy procedures at Cleveland Clinic Florida.
Sampling Method: Probability Sample
Enrollment: 449 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Schneider, M.D., Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Split Dose Colonoscopy Preparation: Esophagogastroduodenoscopy and colonoscopy - split dose - ½ evening before and ½ early AM (4L volume or 2L volume bowel preparation)
  Esophagogastroduodenoscopy and colonoscopy: Patients undergoing a combined EGD (esophagogastroduodenoscopy) and a colonoscopy.
- Evening Before Colonoscopy Preparation: Esophagogastroduodenoscopy and colonoscopy - Evening before (4L, 2L or miralax bowel preparation)
  Esophagogastroduodenoscopy and colonoscopy: Patients undergoing a combined EGD (esophagogastroduodenoscopy) and a colonoscopy.
- Same Day Prep Colonoscopy Preparation: Esophagogastroduodenoscopy and colonoscopy - Same day prep (4L volume or 2L volume or Miralax bowel preparation)
  Esophagogastroduodenoscopy and colonoscopy: Patients undergoing a combined EGD (esophagogastroduodenoscopy) and a colonoscopy.
Period: Overall Study
Arm/Group | Split Dose Colonoscopy Preparation | Evening Before Colonoscopy Preparation | Same Day Prep Colonoscopy Preparation
Started | 21 | 187 | 241
Completed | 21 | 187 | 241
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Split Dose Colonoscopy Preparation | Evening Before Colonoscopy Preparation | Same Day Prep Colonoscopy Preparation | Total
Number analyzed (Participants) | 21 | 187 | 241 | 449
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (13) | 56 (11) | 56 (12) | 56 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 116 | 131 | 258
  Male | 10 | 71 | 110 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 62 | 73 | 140
  Not Hispanic or Latino | 16 | 121 | 160 | 297
  Unknown or Not Reported | 0 | 4 | 8 | 12
Region of Enrollment [Number; unit: participants]
  United States | 21 | 187 | 241 | 449
Diabetes Mellitus [Number; unit: participants] | 5 | 17 | 19 | 41
Constipation [Number; unit: participants] | 3 | 19 | 12 | 34
PPI/H2 Blocker [Number; unit: participants] | 9 | 98 | 117 | 224
Drugs affecting GI motility [Number; unit: participants] | 10 | 94 | 98 | 202
Volume of preparation: 4L [Number; unit: participants] | 21 | 101 | 155 | 277
Last ingestion of solids (hours) [Mean (Standard Deviation); unit: hours] | 35.5 (8.7) | 37.3 (9.8) | 39.4 (9.6) | 38.4 (9.7)
Last ingestion of clear liquids (hours) [Mean (Standard Deviation); unit: hours] | 5.4 (1.9) | 10.3 (4.6) | 5.8 (2.4) | 7.7 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Residual Gastric Volumes of Different Bowel Preparation Regimens
Description: The residual gastric volume for the patients undergoing a combined esophagogastroduodenoscopy and colonoscopy will be measured and compared among the groups taking different bowel preparations.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Split Dose Colonoscopy Preparation | Evening Before Colonoscopy Preparation | Same Day Prep Colonoscopy Preparation
Number analyzed (Participants) | 21 | 187 | 241
mL | 19 (22) | 16 (16) | 18 (20)

2. Secondary Outcome: pH of Gastric Fluid of Different Bowel Preparation Regimens
Description: The pH of gastric fluid for the patients undergoing a combined esophagogastroduodenoscopy and colonoscopy will be measured and compared among the groups taking different bowel preparations.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Split Dose Colonoscopy Preparation | Evening Before Colonoscopy Preparation | Same Day Prep Colonoscopy Preparation
Number analyzed (Participants) | 21 | 187 | 241
pH | 2.1 (1.5) | 2.5 (1.4) | 2.5 (3)

3. Secondary Outcome: Procedure Complications (Decrease in Oxygen Saturation)
Description: The patients will be evaluated for complications namely decrease in oxygen saturation during the procedure (Esophagogastroduodenoscopy and colonoscopy) in three groups.
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Split Dose Colonoscopy Preparation | Evening Before Colonoscopy Preparation | Same Day Prep Colonoscopy Preparation
Number analyzed (Participants) | 21 | 187 | 241
participants | 1 | 6 | 11

ADVERSE EVENTS:
Arm/Group | Split Dose Colonoscopy Preparation | Evening Before Colonoscopy Preparation | Same Day Prep Colonoscopy Preparation
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/187 | 0/241
Other Adverse Events (participants affected / at risk) | 0/21 | 0/187 | 0/241

LIMITATIONS AND CAVEATS:
The patients were not randomized to the two groups. Endoscopists were not blinded to the fact that patients were in the study but were unaware of the preparation type.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes